CLINICAL TRIAL: NCT01720277
Title: High Dose Influenza Vaccination and Morbidity and Mortality in U.S. Nursing Homes - A Pilot Evaluation
Brief Title: High Dose Influenza Vaccine in Nursing Home - Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insight Therapeutics, LLC (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Stefan Gravenstein, MD, MPH, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRC75-HD Nursing Home Pilot
Record Dates: First submitted 2012-10-15; First posted 2012-11-02 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Influenza
Keywords: Randomized Controlled Trial; Influenza; Influenza vaccine; Flu Vaccine; Fluzone; HD Fluzone; Nursing Homes; Hospitalization; Mortality; Health Care worker vaccination; ADL decline; Pilot; Effectiveness
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HD Fluzone Vaccine (Experimental): NH facilities randomized to receive high dose trivalent influenza vaccine (HD Fluzone) for the residents.
  Interventions: Biological: HD Fluzone Vaccine
- SD Fluzone Vaccine (Active Comparator): NH facilities randomized to standard dose trivalent influenza vaccine (SD Fluzone) for the residents.
  Interventions: Biological: SD Fluzone Vaccine

INTERVENTIONS:
Biological: HD Fluzone Vaccine — Nursing home residents over 65 years are allocated to receive high dose trivalent vaccine. Residents under 65 years are provided standard dose trivalent vaccine (TIV).
  Other Names: Fluzone High Dose influenza vaccine
  Arms: HD Fluzone Vaccine
Biological: SD Fluzone Vaccine — Nursing home residents are allocated to receive standard trivalent vaccine (TIV).
  Other Names: Fluzone influenza vaccine
  Arms: SD Fluzone Vaccine

SUMMARY:
The purpose of this pilot evaluation is to help determine the feasibility and power needed to prospectively evaluate relative effectiveness of high-dose influenza vaccine in preventing influenza mortality and hospitalization in a nursing home population in the U.S., compared to the standard-dose influenza vaccine.

DETAILED DESCRIPTION:
Influenza remains the most common preventable respiratory viral infection of older adults. Older adults incur more than 90% of the disease burden, and those residing in nursing homes are the most affected subset given their immune senescence, multi-morbidity, and close living quarters. Each year, the majority of influenza-related hospitalizations occur during the period with the greatest influenza activity.

Influenza vaccination has been associated with reduced hospitalization, strokes, heart attacks and death in non-institutional older adult populations, but the benefit of influenza vaccine for the oldest population has been questioned. The new high-dose influenza vaccine is considerably more immunogenic in older adults, and has recently been approved for use in individuals aged 65 years and older. No clinical data yet confirm whether the improved immunogenicity translates into added clinical benefit, such as further reduction in hospitalization or death. Estimating the benefit of influenza vaccination among older adults in long-term care settings using randomized controlled trials requires extensive effort and is costly. Instead, a pragmatic RCT in a nursing home population has several advantages as a model for comparing therapeutic approaches.

This clinical trial aims to test the feasibility of our protocol for a subsequent larger study. We aim to demonstrate that we can recruit and enroll facilities; randomly assign and coordinate vaccine delivery; collect data; conduct site audits for data validation; create outcomes using multiple data sources; and conduct analyses.

ELIGIBILITY:
Inclusion Criteria:

* Long-term care facilities in one of the 122 cities that serve as Center for Disease Control and Prevention (CDC) surveillance sites

Exclusion Criteria:

* Facilities already systematically administering HD vaccine to their residents
* Facilities for whom over half the residents are on Medicare (short-stay)
* Facilities in which over half the residents are on Medicare Part A (SNF)
* Facilities having fewer than 50 long-stay residents
* Hospital-based facilities
* Facilities with more than 20% of the population under age 65
* Facilities with mandated (employment-dependent) seasonal influenza vaccination
* Facilities not submitting MDS data

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2957 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gravenstein, MD, MPH, Principal Investigator — Case Western Reserve University; Ed Davidson, PharmD, MPH, Principal Investigator — Insight Therapeutics, LLC; Vincent Mor, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Brown Univeristy, Providence, Rhode Island
  - Insight Therapeutics, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Bridges CB, Cox NJ, Fukuda K. Influenza-associated hospitalizations in the United States. JAMA. 2004 Sep 15;292(11):1333-40. doi: 10.1001/jama.292.11.1333. PMID 15367555
- [Background] Hayward AC, Harling R, Wetten S, Johnson AM, Munro S, Smedley J, Murad S, Watson JM. Effectiveness of an influenza vaccine programme for care home staff to prevent death, morbidity, and health service use among residents: cluster randomised controlled trial. BMJ. 2006 Dec 16;333(7581):1241. doi: 10.1136/bmj.39010.581354.55. Epub 2006 Dec 1. PMID 17142257
- [Background] Deguchi Y, Nishimura K. Efficacy of Influenza Vaccine in Elderly Persons in Welfare Nursing Homes: Reduction in Risks of Mortality and Morbidity During an Influenza A (H3N2) Epidemic. J Gerontol A Biol Sci Med Sci. 2001 Jun;56(6):M391-4. doi: 10.1093/gerona/56.6.m391. PMID 11382801
- [Background] Gozalo PL, Pop-Vicas A, Feng Z, Gravenstein S, Mor V. Effect of influenza on functional decline. J Am Geriatr Soc. 2012 Jul;60(7):1260-7. doi: 10.1111/j.1532-5415.2012.04048.x. Epub 2012 Jun 21. PMID 22724499
- [Background] Barker WH, Borisute H, Cox C. A study of the impact of influenza on the functional status of frail older people. Arch Intern Med. 1998 Mar 23;158(6):645-50. doi: 10.1001/archinte.158.6.645. PMID 9521230
- [Background] Jackson LA, Jackson ML, Nelson JC, Neuzil KM, Weiss NS. Evidence of bias in estimates of influenza vaccine effectiveness in seniors. Int J Epidemiol. 2006 Apr;35(2):337-44. doi: 10.1093/ije/dyi274. Epub 2005 Dec 20. PMID 16368725
- [Background] Simonsen L, Viboud C, Taylor R. Influenza vaccination in elderly people. Lancet. 2005 Dec 17;366(9503):2086. doi: 10.1016/S0140-6736(05)67884-1. No abstract available. PMID 16360785
- [Background] Fiore AE, Shay DK, Haber P, Iskander JK, Uyeki TM, Mootrey G, Bresee JS, Cox NJ; Advisory Committee on Immunization Practices (ACIP), Centers for Disease Control and Prevention (CDC). Prevention and control of influenza. Recommendations of the Advisory Committee on Immunization Practices (ACIP), 2007. MMWR Recomm Rep. 2007 Jul 13;56(RR-6):1-54. PMID 17625497
- [Background] Kingston BJ, Wright CV Jr. Influenza in the nursing home. Am Fam Physician. 2002 Jan 1;65(1):75-8, 72. PMID 11804444
- [Background] Menec VH, Black C, MacWilliam L, Aoki FY. The impact of influenza-associated respiratory illnesses on hospitalizations, physician visits, emergency room visits, and mortality. Can J Public Health. 2003 Jan-Feb;94(1):59-63. doi: 10.1007/BF03405054. PMID 12583681
- [Background] Mor V, Intrator O, Unruh MA, Cai S. Temporal and Geographic variation in the validity and internal consistency of the Nursing Home Resident Assessment Minimum Data Set 2.0. BMC Health Serv Res. 2011 Apr 15;11:78. doi: 10.1186/1472-6963-11-78. PMID 21496257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cluster--We included nursing homes (NHs) within 50 miles of a CDC surveillance. We identified and contacted individual facilities and organizations. Each recruited NH completed a site feasibility form and was notified of its eligibility based on the exclusion criteria.
  Subject--Eligible nursing home residents in each participating facility.
Units Other Than Participants: nursing home
Groups:
- High-Dose Vaccine for Residents: NH facilities randomized to receive high dose trivalent influenza vaccine (High-dose Fluzone) for the residents.
- Standard-dose for Residents: NH facilities randomized to receive free standard-dose trivalent influenza vaccine (Fluzone) for nursing home residents.
Period: Overall Study
Arm/Group | High-Dose Vaccine for Residents | Standard-dose for Residents
Started | 1461; 20 nursing home | 1496; 19 nursing home
Completed | 958; 20 nursing home (intent-to-treat approach) | 938; 19 nursing home (intent-to-treat approach)
Not Completed | 503; 0 nursing home | 558; 0 nursing home

BASELINE CHARACTERISTICS:
Population: Characteristics of participating facilities that met our inclusion criteria and were randomized.
  Residents in each participating facility were offered influenza vaccine according to the randomization.
Units Other Than Participants: nursing homes
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Dose Vaccine for Residents | Standard-dose for Residents | Total
Number analyzed (Participants) | 1461 | 1496 | 2957
Number analyzed (nursing homes) | 20 | 19 | 39
Age, Customized [Mean (Standard Deviation); unit: years]
  Average age | 84.5 (8.4) | 83.4 (8.7) | 84.0 (8.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Percent of female nursing home residents | 1094 | 1113 | 2207
Number of residents per nursing home [Mean (Standard Deviation); unit: participants] | 108 (49) | 124 (54) | 116 (51)
Percent of residents who are long-stay [Mean (Standard Deviation); unit: percent] | 88.0 (6.5) | 86.5 (12.1) | 87.2 (9.7)
Number of long-stay residents who are over 65 years of age [Mean (Standard Deviation); unit: participants] | 78 (37) | 78 (44) | 78 (40)
Percent of residents with Medicaid as payer [Mean (Standard Deviation); unit: percent] | 62.5 (12.8) | 62.9 (17.4) | 62.7 (15.0)
Percent of residents in for-profit nursing facilities [Mean (Standard Deviation); unit: percent] | 70.0 (47.0) | 73.6 (45.2) | 71.8 (45.6)
Number of nursing facilities that are part of a chain [Number; unit: nursing homes] | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Total All-cause Hospitalizations
Description: The primary outcome will establish our methodology for measuring all-cause hospitalizations using the Minimum Data Set (MDS).
Time Frame: 1 year
Population: We identified long-stay nursing home residents and evaluated outcomes (e.g. hospitalizations, functional status).
Measure: Number; unit: events
Arm/Group | High-Dose Vaccine for Residents | Standard-dose for Residents
Number analyzed (Participants) | 1461 | 1496
events | 197 | 301

2. Secondary Outcome: Change in Residents' Functional Status
Description: The secondary outcome will establish our methodology for measuring change in functional status of nursing home residents using Activities of Daily Living (ADL) data in the Minimum Data Set (MDS). A change in functional status is defined as a decline in physical functioning by at least 4 points on the 28-point ADL scale.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | HD Fluzone Vaccine | SD Fluzone Vaccine
Number analyzed (Participants) | 1461 | 1496
Participants | 196 | 206

3. Other Pre Specified Outcome: Recruit, Enroll, and Randomize Nursing Homes Per Calculated Sample Size
Description: This outcome evaluates our ability to recruit and enroll nursing facilities that meet our inclusion and exclusion criteria, and ensure nursing home residents receive either high-dose or standard-dose influenza vaccine
Time Frame: 1 year
Population: Nursing home facilities randomized to receive high dose or standard dose vaccine.
Measure: Number; unit: Nursing Homes
Units Other Than Participants: Nursing Homes
Arm/Group | HD Fluzone Vaccine | SD Fluzone Vaccine
Number analyzed (Participants) | 20 | 19
Number analyzed (Nursing Homes) | 20 | 19
Nursing Homes | 20 | 19

ADVERSE EVENTS:
Time Frame: The study did not collect adverse events.
Description: The study did not collect adverse events.
Arm/Group | High-Dose Vaccine for Residents | Standard-dose for Residents
All-Cause Mortality (participants affected / at risk) | 249/1461 | 274/1496
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No